CLINICAL TRIAL: NCT04375501
Title: The Effects of Coronavirus on Perioperative Morbidity and Mortality in a High-risk Population: A Multicentre Cohort Study
Brief Title: A Study of Outcomes in Patients With Fractured Neck of Femur During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: University College London Hospitals (Other); Barking, Havering and Redbridge University Hospitals NHS Trust (Other); Mid and South Essex NHS Foundation Trust (Other); Frimley Park Hospital NHS Trust (Other); The Hillingdon Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Elliot Onochie, Author and Investigator, Barts & The London NHS Trust
Other Study IDs: 284104
Record Dates: First submitted 2020-05-04; First posted 2020-05-05 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Femoral Neck Fractures; SARS-CoV 2
Keywords: COVID-19; Coronavirus; Neck of femur; Morbidity; Mortality; Prognosis
MeSH Terms: conditions — Femoral Neck Fractures; COVID-19; Coronavirus Infections | interventions — Hemiarthroplasty; Arthroplasty, Replacement, Hip; Fracture Fixation, Intramedullary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 positive: All patients admitted with fractured neck of femur during specified time period testing POSITIVE for COVID-19
  Interventions: Other: Surgery: Dynamic Hip Screw, hemiarthroplasty, hip replacement, intramedullary nail
- COVID-19 negative: All patients admitted with fractured neck of femur during specified time period testing NEGATIVE for COVID-19
  Interventions: Other: Surgery: Dynamic Hip Screw, hemiarthroplasty, hip replacement, intramedullary nail

INTERVENTIONS:
Other: Surgery: Dynamic Hip Screw, hemiarthroplasty, hip replacement, intramedullary nail — If fit for anaesthesia patients may undergo relevant procedure for fractured neck of femur as per NICE guidelines within limitations of resources as defined by BOAST

SUMMARY:
In early 2020 the evolving COVID-19 Pandemic provided the world and medical community with a generational challenge. As a novel disease, countries were left with strategic decisions and many went into social lockdown. Initial resources and research were directed at upscaling internal medicine and intensive care services, understanding the disease pathophysiology, and testing treatments. It soon became evident that COVID-19 had multi-system effects at it's worst. In orthopaedics one of the most vulnerable groups to COVID-19 were the elderly, specifically those who suffered fractured neck of femur at this time. More literature is needed urgently if we are to understand and mitigate the negative impacts in this group of patients. This observational study assesses the early morbidity and mortality of patients with this diagnosis during the evolving COVID-19 Pandemic.

DETAILED DESCRIPTION:
Many elderly patients admitted to hospitals during the evolving COVID-19 pandemic after falls or being generally unwell, were considered to have a possible diagnosis of COVID-19. This was extremely relevant to the subgroup of patients who suffered from fractured neck of femurs during this time, with most of them elderly, frail, and more likely to have multiple co-morbidities. COVID-19 was considered a precipitating factor for falls, but also anecdotally, an indicator of potentially poor recovery and rehabilitation.

With regards to orthopaedic and trauma surgery, a limited amount of literature is available pertaining to COVID-19 and specifically it's potential effects on patient outcomes in patients requiring surgery.

We performed a multi centre observational study across London, United Kingdom, looking at the demographics and details of patients admitted with fractured neck of femur during the evolving pandemic. All data collected was non identifiable. Data was also collected as to the COVID-19 status of these patients, either positive or negative. Data was analysed to assess the morbidity and mortality of this patient group and search for any prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Fractured neck of femur
* Received operative intervention for fractured neck of femur

Exclusion Criteria:

* open fracture
* fracture of femoral shaft
* periprosthetic fracture
* revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted February 1st 2020 to April 15th 2020 with fractured neck of femur
Sampling Method: Non-Probability Sample
Enrollment: 442 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 day
  Death
Morbidity | 30 day
  Morbidity

SECONDARY OUTCOMES:
Discharge | 30 day
  Discharge to home, rehabilitation or community setting

CONTACTS AND LOCATIONS:
Overall Officials: Babar Kayani, MBBS, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared